CLINICAL TRIAL: NCT00399555
Title: Neurodevelopmental Outcomes in Hypoplastic Left Heart Syndrome-Correlation With Cerebral Non-invasive Infrared Spectroscopy (NIRS)
Brief Title: Neurodevelopmental Outcomes in Hypoplastic Left Heart Syndrome
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Professor of Pediatrics, Emory University
Other Study IDs: IRB00000275
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Heart Disease
Keywords: Single Ventricle; Hypoplastic Left Heart; Developmental
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One: Patients with HLHS that have had surgical palliation with the Norwood procedure (Stage I palliation) at Children's Healthcare of Atlanta after January 1, 2001. These patients must be between the ages of 2.5 years and 6 years of age.

SUMMARY:
There have been many improvements in the care of children with hypoplastic left heart syndrome (HLHS). This has helped these children survive longer. Because these children now live longer, researchers are recognizing developmental disabilities (the children are behind in their thinking or physical activity) in children with hypoplastic left heart syndrome. The purpose of this research study is to help the investigators learn more about developmental disabilities in children with hypoplastic left heart syndrome.

During the time of your child's first surgery for hypoplastic left heart syndrome, a monitor was placed on your child's forehead to measure the oxygen levels in the brain. This monitor is called Near Infrared Spectrometry (NIRS). The researchers involved in this study want to know if oxygen levels in the blood vessels of the brain have any effect on developmental disabilities later in life in children with hypoplastic left heart syndrome. The researchers plan to enroll 60 research subjects.

DETAILED DESCRIPTION:
Our study is a cross-sectional, descriptive study to evaluate the developmental outcome for school-age children with HLHS. The general approach of the proposed research is confirmatory study/hypothesis testing. The hypothesis (neurodevelopmental outcome of children with HLHS is inversely correlated with cerebral oximetry values as measured by NIRS in the 48 hours following the Norwood operation) was formulated based on a meticulous review of the literature, which clearly demonstrates a substantial prevalence of neurodevelopmental deficits in children with HLHS who have undergone surgical palliation. The methodologies for measuring developmental outcome are highly reproducible and have been validated in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Hypoplastic left heart syndrome is defined as normal segmental anatomy with mitral and/or aortic atresia or stenosis and a left ventricle too small to sustain the systemic circulation
2. Ages 2.5 to 6 years old
3. Surgical palliation with the Norwood procedure (Stage I palliation) at Children's Healthcare of Atlanta after January 1, 2001

Exclusion Criteria:

1. Primary language in the home is not English
2. Named genetic syndrome associated with profound developmental delay, such as DiGeorge Syndrome

Ages: 29 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 2.5 to 6 years old who have hypoplastic left heart syndrome with surgical palliation and near infrared spectrometry monitoring during the Stage I Norwood procedure.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To describe the developmental outcome of school-age children with HLHS who have undergone the Norwood procedure at our institution after January 1, 2001 | Ages 2.5 years to 6 years

SECONDARY OUTCOMES:
Determine whether there is a correlation between cerebral oxygen levels as measured by NIRS and subsequent developmental outcome | NIRS measurement 48 hours after Norwood procedure and developemental outcome by 2.5-6 years of age

CONTACTS AND LOCATIONS:
Overall Officials: William Mahle, MD, Study Director — Sibley Heart Center/Emory Universtiy School of Medicine
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States